

CLINICAL TRIAL PROTOCOL NUMBER: APX-23-02

Measuring Renuvion Soft Tissue Contraction Using Ultrasound

SPONSOR: APYX MEDICAL

FUNDED BY: APYX MEDICAL

DATE: MAY 23, 2023

DRAFT OR VERSION: 1.1

CONFIDENTIAL - PROPRIETARY INFORMATION

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



## SPONSOR STATEMENT AND SIGNATURE PAGE

Company Name: Apyx Medical
Address: 5115 Ulmerton Rd.
Clearwater, FL 33760

800.537.2790

Study Device: Apyx Plasma RF

Protocol Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound

Protocol Number: APX-23-02

Telephone:

The investigation will be conducted in compliance with the clinical investigation plan (CIP), GCP, EN ISO 14155, the Declaration of Helsinki, and regulatory authority requirements.

Apyx Medical (hereinafter "Study Sponsor") maintains responsibility for the ongoing safety of this clinical trial involving the evaluation of the Renuvion system. Study Sponsor will promptly notify all investigators, the responsible IRB(s), and the regulatory authorities of any findings from ongoing trial monitoring activities that could adversely affect the safety of subjects, impact the conduct of the clinical study, or alter the IRB's approval to continue the study, specifically within 5 working days of making an Unanticipated Adverse Device Effect (UADE) determination or 15 working days after first receiving notice of the UADE, within 10 days for Serious Adverse Event reports, and at least annually for routine reports. In the event that participant safety could be directly affected by study results after the study has ended, Study Sponsor will notify all investigators of these results to enable investigators to consider informing participants as soon as possible or at least within one year of study closure.

The following individuals are responsible for the content of the CIP:

| Emily Hughes | Date |
|--------------------------------------------------------|------|
| Sr. Manager, Clinical Affairs | |
| Kari Larson | Date |
| Sr. Director, Clinical Affairs | |
| Shawn Roman | Date |
| Vice-President, R&D | |
| Lisa Graney | Date |
| Vice-President, Quality Assurance & Regulatory Affairs | |

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



# INVESTIGATOR AGREEMENT/STATEMENT OF COMPLIANCE

I have thoroughly read and reviewed this clinical investigation plan (CIP) and hereby agree to participate in this clinical trial sponsored by Study Sponsor. I agree to conduct this investigation according to the requirements of the CIP provided by the Study Sponsor and in accordance with Good Clinical Practice (GCP) as required by EN ISO 14155, the Declaration of Helsinki, Investigational Device Exemption (21 CFR Part 812), Protection of Human Subjects (45 CFR Part 46), and other applicable FDA regulations, and regulations of other relevant regulatory authorities and conditions imposed by the reviewing Institutional Review Board (IRB) or Ethics Committee (EC). I agree that no deviation from, or changes to the CIP will take place without prior agreement from the sponsor and documented approval from the IRB, except where necessary to eliminate an immediate hazard(s) to the trial participants. I agree to ensure that appropriate informed consent is obtained from all subjects prior to inclusion in this study. I also agree to supervise all testing of the device involving human subjects, and to report to the Study Sponsor, within 24 hours, any adverse event that is serious, whether considered treatment-related or not. I am aware that the Study Sponsor reserves the right to discontinue this investigation at any time.

I understand that this investigation will be monitored by the Study Sponsor and/or a designee employed by the Study Sponsor. This monitoring will involve periodic inspection of my investigational site and ongoing review of the data that is submitted by me to the Study Sponsor.

All study data will be entered into the EDC and a PDF of the paper CRF will be uploaded to the EDC within 3 days after the study visit.

I am also aware that I may be inspected by a representative of the relevant regulatory authorities, including the United States Food and Drug Administration, to verify compliance with applicable regulations related to clinical research on human subjects.

My current curriculum vitae and the curriculum vitae of physicians/licensed practitioners at this institution who will participate as co-investigators/sub-investigators in this study will be provided to the Study Sponsor. The curriculum vitae will include the extent and type of our relevant experience with pertinent dates and locations. All personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I certify that I have not been involved in an investigation that was terminated for non-compliance at the insistence of the Study Sponsor, the IRB or EC, or other regulatory authorities. I agree to provide the Study Sponsor sufficient, accurate financial disclosure information. I also agree to update financial disclosure information if any relevant changes occur during the investigation and for one year following the completion of the study.

I understand that this CIP and the trial results are confidential, and I agree not to disclose any such information to any person other than a representative of the Study Sponsor or the relevant competent authorities without the prior written consent of the Study Sponsor.

| Accepted by: | | |
|-------------------------------------|-----------------------------|----------|
| Co-Principal Investigator Signature | Principal Investigator Name | Date |
| Co-Principal-Investigator Signature | Co-Investigator Name | <br>Date |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



**Revision No:** 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|---|---|
| CRF | Case Report Form |
| CRO | Clinical Research Organization |
| DCF | Data Clarification Form |
| DRM | Data Review Meeting |
| ESU | Electrosurgical Generator Unit |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| GAIS | Global Aesthetic Improvement Scale |
| GCP | Good Clinical Practice |
| ICH | International Conference for Harmonization of Technical Requirements of Pharmaceuticals for Human Use |
| IFU | Instructions for Use |
| IPR | Independent Photographic Reviewer |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| NRS | Numeric Rating Scale |
| NSAID | Non-steroidal Anti-Inflammatory Drug |
| PP | Per Protocol |
| PPS | Per Protocol Set |
| RF | Radiofrequency |
| SAE | Serious Adverse Event |
| SAL | Suction-Assisted Liposuction |
| UADE | Unanticipated Adverse Device Effect |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

# **PROTOCOL SYNOPSIS**

| Protocol Title: | Measuring Renuvion Soft Tissue Contraction Using Ultrasound |
|---|---|
| Investigational Device: | The Renuvion Generator (K192867) is indicated for delivery of radiofrequency energy and/or helium plasma to cut, coagulate and ablate soft tissue during open and laparoscopic surgical procedures. The Renuvion APR Handpiece (K223262) is intended for the delivery of radiofrequency energy and/or helium plasma where coagulation/contraction of soft tissue is needed. Soft tissue includes subcutaneous tissue. The Renuvion® APR Handpiece is indicated for use in subcutaneous dermatological and aesthetic procedures to improve the appearance of lax (loose) skin in the neck and submental region. The Renuvion® APR Handpiece is intended to be used with compatible electrosurgical generators owned by Apyx Medical. The Apyx One Console (K221830) is indicated for delivery of radiofrequency energy and/or helium plasma to cut, coagulate and ablate soft tissue during open and laparoscopic surgical procedures. The helium plasma portion of the generator can be used only with dedicated Renuvion/J-Plasma handpieces. |
| | Together, the Renuvion Generator and Handpiece are referred to as the Renuvion APR System. |
| Development Phase: | Post-Marketing |
| Study Purpose: | The purpose of this study is to quantitatively measure the amount of soft tissue contraction produced by the delivery of Renuvion helium plasma energy to the subcutaneous connective tissue. |
| Brief Study Overview: | This is a prospective, single-center, non-randomized study of up to 5 subjects who are receiving treatment with the Renuvion APR system following power-assisted liposuction in the abdomen per investigator standard of care. Subjects may also have other body areas treated at the same time. Demographic information, medical history, and procedure details will be documented. Pre- and post-procedure care are per investigator standard of care and documented. Video may be taken during the procedure. |
| | Ultrasound images of soft tissue contraction will be taken on abdomen prior to and during the procedure. Measurements of contraction will be calculated from the ultrasound images by an ultrasonographer. At baseline, photographs will be taken of the treatment areas. Surface area measurements will be taken of each treatment area prior to study treatment. |
| | Post-procedure care will be as per investigator standard of care and documented. All adverse events and expected treatment effects will be documented. |
| | Follow-up photographs and ultrasound images will be captured at D30, D45, D60, D90, D180, D270, & D365. |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



| | An interim analysis of data will be completed following study treatments and following each follow-up visit (D30, D45, D60, D90, D180, D270); a final report will provide comprehensive study results through D365. |
|---|---|
| Number of Sites Enrolling Participants: | Subjects will be recruited from a single (1) US site. |
| Sample Size: | Up to 5 treated subjects; subjects enrolled may be greater than subjects treated. |
| Subject Population: | Healthy, female and male adult subjects, ages 18 – 65 years old who meet the inclusion/exclusion criteria. |
| Inclusion Criteria: | <ul> <li>Patients who are scheduled for a procedure involving the use of Renuvion for the contraction of subcutaneous soft tissue. Patients undergoing procedures involving Renuvion alone and/or Renuvion following liposuction will be included.</li> <li>Patients who have acceptable cardiopulmonary health for outpatient surgery.</li> <li>Willing and able to comply with protocol requirements, including obtaining study-required images/photos and assessments, and returning for follow-up visits.</li> <li>Willing to release rights for the use of study photos, including in potential publication.</li> <li>Able to communicate with the site via video and/or photographs, in the event of a virtual follow-up visit.</li> <li>Able to read, understand, sign and date the informed consent document (English only).</li> </ul> |
| Exclusion Criteria: | <ul> <li>BMI of greater than 35.</li> <li>Diabetes mellitus with A1C score &gt;7.</li> <li>Active cigarette smokers or nicotine vape users.</li> <li>History of connective tissue disease (Ehlers Danlos, Cutis Laxa, Pseudoxanthoma Elasticum, Marfan's, etc.)</li> <li>Patients who, in the opinion of the investigator, is not an appropriate candidate for the study.</li> </ul> |
| | <ul> <li>Patients requiring a concomitant procedure in the Renuvion treatment area that<br/>could impact the ultrasound measurements or the effectiveness results.</li> </ul> |
| Primary Outcome<br>Measures: | <ul> <li>Analysis of contraction measured by an ultrasonographer and then analyzed as follows:</li> <li>Quantify the amount of intra-operative contraction produced by liposuction.</li> <li>Quantify the amount of intra-operative contraction produced by each pass of Renuvion.</li> <li>Determine if amount of intra-operative contraction produced by Renuvion begins to level off (reach a point of diminishing return).</li> <li>Determine how the amount of intra-operative contraction varies based on the initial length at baseline.</li> <li>Correlate the amount of intra-operative contraction to energy delivered.</li> <li>Determine how the amount of contraction changes over time.</li> <li>Correlate the amount of contraction to GAIS and PSQ.</li> <li>Correlate the amount of contraction or energy delivered to AEs.</li> <li>Correlate the amount of contraction to IPR review.</li> </ul> |
| Additional Outcome<br>Measures: | 1. Improvement in appearance of skin laxity in the treatment area assessed by selection of the correct post-treatment image as determined by a masked, qualitative |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



| | <ol> <li>assessment of photographs by blinded independent reviewers at 90-days, 180-days, 270-days, and 365-days post-treatment compared to baseline.</li> <li>The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a PGAIS assessing overall aesthetic improvement in the treatment area at day 60, 90, 180, 270, and 365 post-treatment.</li> <li>The subject will complete a SGAIS assessing overall aesthetic improvement in the treatment area at day 60, 90, 180, 270, and 365 post-treatment.</li> <li>The subject will complete a Patient Satisfaction Questionnaire (PSQ) at the 180-, 270-and 365-day follow-up visits.</li> <li>Analysis of energy delivered per surface area and per volume of tissue.</li> </ol> |
|---|---|
| Safety Variables: | <ul> <li>Prior to treatment, the subject's medical history will be reviewed, a urine pregnancy test will be performed (if applicable), and a physical examination will be conducted.</li> <li>Following study treatment and at each subsequent visit, the subject will be queried about adverse events, expected treatment effects, and changes in concomitant medications, and the treatment area will be visually examined.</li> <li>Analysis of adverse events through the D365 post-treatment visit.</li> </ul> |
| Study Duration: | The duration from when the study opens to enrollment until completion of data analyses is anticipated to be 16 months. |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Protocol Number: APX-23-02

Effective Date: May 23, 2023

**Revision No: 1.1** 

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

# TABLE OF CONTENTS

| Spons | or Statement and Signature Page | |
|---|---|---|
| Invest | gator Agreement/Statement of Compliance | ŝ |
| List of | Abbreviations | 4 |
| | ol Synopsis | |
| | KEY ROLES | |
| 1.1 | Internal Responsibilities | |
| 1.2 | External Responsibilities | |
| 2. | NTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE | 13 |
| 2.1 | Background Information & Rationale | 13 |
| 2.1 | | |
| 2.1 | · | |
| 2.2 | Potential Risks and Benefits | 1 |
| 2.2 | .1 Potential Risks | 1 |
| 2.2 | .2 Potential Benefits | 18 |
| <b>3.</b> | STUDY PURPOSE | 19 |
| 4. | STUDY DESIGN AND ENDPOINTS | 19 |
| 4.1 | Description of the Study Design | 19 |
| 4.2 | Duration of Study | 19 |
| 4.3 | Study Endpoints | 19 |
| 4.3 | .1 Primary Effectiveness Endpoint | 19 |
| 4.3 | .2 Safety Variables | 20 |
| 4.3 | .3 Additional Outcome Measures | 20 |
| 4.3 | .4 Evaluation Tools | 20 |
| <b>5.</b> . | SUBJECT ENROLLMENT AND WITHDRAWAL | 22 |
| 5.1 | Study Population | 22 |
| 5.1 | | |
| 5.1 | .2 Pre-treatment Recruiting/Screening | 23 |
| 5.2 | Inclusion Criteria | 2 |
| 5.3 | Exclusion Criteria | 24 |



**Revision No:** 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

| 5.4 | Strator | es for Recruitment and Retention | 2/ |
|---|---|---|---|
| _ | | | |
| 5.5 | = | ant Withdrawal or Termination | |
| | | asons for Withdrawal or Termination | |
| 5 | .5.2 Ha | ndling of Withdrawals or Termination | 24 |
| 5.6 | Premate | ure Termination or Suspension of the Study or a Study Site | 25 |
| <i>6.</i> | STUDY D | PEVICE | 25 |
| 6.1 | Dackagi | ng & Storage | 20 |
| | _ | | |
| 6.2 | Accoun | tability | 26 |
| 6.3 | Device I | Malfunction/Observation | 26 |
| <b>7.</b> | STUDY P | ROCEDURES AND SCHEDULE | 26 |
| 7.1 | Pre-Pro | cedure | 76 |
| 7.2 | Study P | rocedure | 26 |
| 7.3 | Follow- | up Procedures | 27 |
| | | iately Post-Procedure | |
| 7 | .3.2 Follow- | up Visits & Subject Contact outside of Follow-up Visits | 27 |
| 7.4 | Subject | Randomization and Treatment Group Assignment | 28 |
| 7.5 | Study S | chedule | 28 |
| 7 | .5.1 Scr | eening | 28 |
| 7 | .5.2 Bas | seline Assessment | 28 |
| 7 | .5.3 Tre | eatment Visit | 29 |
| 7 | .5.4 Fol | low-up | 29 |
| 7 | .5.5 Saf | ety Assessments | 30 |
| 7 | | scheduled Visit | |
| 7 | .5.7 End | d of Study (Completion) | 30 |
| 8. | ASSESSN | IENT OF SAFETY | 3C |
| 8.1 | Specific | ations of Safety Parameters | 30 |
| 8 | .1.1 De | finition of an Expected Treatment Effect (ETE) and an Adverse Event (AE) | 30 |
| 8 | .1.2 De | finition of Serious Adverse Event (SAE) | 31 |
| 8 | .1.3 De | finition of Unanticipated Adverse Device Effects (Events) | 31 |
| 8.2 | Classific | ation of an Event | 32 |
| 8 | .2.1 Sev | erity of Event | 32 |
| 8 | .2.2 Rel | ationship to the Investigational Device | 32 |
| 8.3 | Time Pe | riod and Frequency for Event Assessment and Follow-up | 32 |
| 8.4 | Reporti | ng Procedures | 37 |
| | | u | |



**Revision No:** 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

| | 8.4.1 | Adverse Event Reporting | 33 |
|---|---|---|---|
| | 8.4.2 | Serious Adverse Event Reporting | 33 |
| | 8.4.3 | Unanticipated Adverse Device Effect Reporting | 34 |
| | 8.4.4 | Reporting of Pregnancy | |
| | 8.4.5 Re | eporting of Deaths | 34 |
| 8. | 5 Stu | udy Halting Rules | 34 |
| 9. | CLIN | IICAL MONITORING | 35 |
| 10. | Stat | istical Methodology | 35 |
| 10 | .1 Sta | atistical and Analytical Plans | 35 |
| 10 | .2 Sa | mple Size | 35 |
| 11. | sou | RCE DOCUMENTS AND ACCESS TO SOURCE DATA/ DOCUMENTS | 35 |
| 12. | QUA | ALITY ASSURANCE AND QUALITY CONTROL | 35 |
| 13. | ETH | ICS/PROTECTION OF HUMAN SUBJECTS | 36 |
| 13 | .1 Etl | nical Standard | 36 |
| 13 | .2 Ins | titutional Review Board | 36 |
| 13 | .3 Pa | rticipant and Data Confidentiality | 36 |
| 14. | DAT | A HANDLING AND RECORD KEEPING | 37 |
| 14 | .1 Da | ta Collection and Management Responsibilities | 37 |
| 14 | .2 Inv | vestigator Records and Reports | 38 |
| | 14.2.1 | Investigator Records | 38 |
| | 14.2.2 | Investigator Reports | 39 |
| 14 | .3 Stu | udy Records Retention | 39 |
| 14 | .4 Pro | otocol Deviations | 40 |
| 14 | .5 Pu | blication and Data Sharing Policy | 40 |
| <i>15</i> . | STU | DY ADMINISTRATION | 40 |
| 15 | .1 St | udy Investigators | 40 |
| 15 | .2 An | nendment Policy | 41 |
| 16. | CON | IFLICT OF INTEREST POLICY | 41 |
| 17. | LITE | RATURE REFERENCES | 42 |
| ATT | АСНМ | ENT A: PATIENT SATISFACTION QUESTIONNAIRE | 44 |



PROTOCOL REVISION LOG....... 45

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



## 1. KEY ROLES

Persons, companies, and/or groups serving in key roles in the conduct or oversight of this clinical trial are listed in **Table 1** and **Table 2**, including sponsor, clinical project manager for the trial, investigator responsible for conducting the trial. Additional details are available in the study specific Project Plan.

### 1.1 Internal Responsibilities

#### **TABLE 1: INTERNAL RESPONSIBILITIES**

| Name | Function | Address |
|---|---|---|
| Apyx Medical | Sponsor | 5115 Ulmerton Road<br>Clearwater, FL |
| Emily Hughes | Sr. Manager, Clinical Affairs | Phone: 731.414.2603<br>Email: Emily.Hughes@apyxmedical.com |
| Kari Larson | Sr. Director, Clinical Affairs | Phone: 801.244.0058<br>Email: Kari.Larson@apyxmedical.com |
| Shawn Roman | VP, R&D and Clinical Affairs | Phone: 904.382.4857<br>Email: Shawn.Roman@apyxmedical.com |

#### 1.2 EXTERNAL RESPONSIBILITIES

The administrative structure for external responsibilities includes, but is not limited to, the participants in **Table 2**:

#### **TABLE 2: EXTERNAL RESPONSIBILITIES**

| Name | Function | Address |
|---|---|---|
| Chris Nichols, MD | Co-Principal Investigator | Pearl Plastic Surgery & Medical Spa |
| | | 145 Lilly Road NE |
| | | Olympia, WA 98501 |
| | | Phone: 360-878-9300 |
| | | Email: cnichols@pearlplasticsurgery.com |
| Dan Albershardt, MD | Co-Principal Investigator & | Pearl Plastic Surgery & Medical Spa |
| , | Ultrasonographer | 145 Lilly Road NE |
| | | Olympia, WA 98501 |
| | | Phone: 360-878-9300 |
| | | Email: doctordan@pearlplasticsurgery.com |
| Castor | EDC | Phone: 628-239-3493 |
| | | Email: ted.mehalic@castoredc.com |
| Dropbox | Secure cloud-based document | N/A |
| | repository for CRF and images | |
| | upload | |

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

# 2. INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

### 2.1 BACKGROUND INFORMATION & RATIONALE

Energy has been applied in some form to tissue since the beginning of recorded history. The practice of applying heat to tissue through the use of cauteries was used for thousands of years as an invaluable method of controlling hemorrhage. Continuous improvement of methods for utilizing the beneficial effects of heat on tissue eventually led to the development of the basic concepts of electrosurgery we know today. In October of 1926, Dr. Harvey Cushing used an electrosurgical unit developed by Dr. William T. Bovie to successfully remove a highly vascularized brain tumor from a patient after previous failed attempts. Today, electrosurgical instruments are used in almost every surgical procedure performed worldwide.<sup>1</sup>

Through this long history, the heat effects of the radiofrequency (RF) alternating current used in electrosurgery on cells and tissue have been well established. Normal body temperature is 37°C and, with normal illness, can increase to 40°C without permanent impact or damage to the cells of our body. However, when the temperature of cells in tissue reaches 50°C, cell death occurs in approximately 6 minutes.<sup>2</sup> When the temperature of cells in tissue reaches 60°C, cell death occurs instantaneously.<sup>3</sup> Between the temperatures of 60°C and just below 100°C, two simultaneous processes occur.<sup>1</sup> The first is protein denaturation leading to coagulation which will be discussed in more detail below. The second is desiccation or dehydration as the cells lose water through the thermally damaged cellular wall. As temperatures rise above 100°C, intracellular water turns to steam and tissue cells begin to vaporize as a result of the massive intracellular expansion that occurs. Finally, at temperatures of 200°C or more, organic molecules are broken down into a process called carbonization. This leaves behind carbon molecules that give a black and/or brown appearance to the tissue.

Understanding these heat effects of RF energy on cells and tissue can allow the predictable changes to be used to accomplish beneficial therapeutic results. Protein denaturation leading to soft tissue coagulation is one of the most versatile and widely utilized tissue effects. Protein denaturation is the process in which hydrothermal bonds (crosslinks) between protein molecules, such as collagen, are instantaneously broken and then quickly reformed as tissue cools. This process leads to the formation of uniform clumps of protein typically called coagulum through a subsequent process known as coagulation. In the process of coagulation, cellular proteins are altered but not destroyed and form protein bonds that create homogenous, gelatinous structures. The resulting tissue effect of coagulation is extremely useful and most commonly used for occluding blood vessels and causing hemostasis.

In addition to causing hemostasis, coagulation results in predictable contraction of soft tissue. Collagen is one of the main proteins found in human skin and connective tissue. The coagulation/denaturation temperature of collagen is conventionally stated to be 66.8°C, although this can vary for different tissue types.<sup>4</sup> Once denatured, collagen rapidly contracts as fibers shrink to one-third of their overall length.<sup>5</sup> This principal of thermally-induced contraction of collagen through denaturation and coagulation of soft tissue is well known in medicine and is used to achieve beneficial results in ophthalmology, orthopedic applications, and the treatment of varicose veins. Once tissue is heated to the appropriate temperature, protein denaturation and collagen contraction occur resulting in a reduction of volume and surface area of the heated tissue. Noninvasive use of RF devices, lasers, and plasma devices have been used for the reduction of facial wrinkles and rhytides caused by thermal-induced collagen/tissue contraction since the mid-1990s.<sup>6-11</sup>

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

Minimally invasive devices that deliver thermal energy in the same subcutaneous tissue planes in which liposuction is performed have achieved the appropriate balance between excisional and non-invasive procedures. Laser-assisted liposuction (LAL) has shown to be effective at producing more skin tightening than suction-assisted liposuction (SAL) alone<sup>18,19</sup>. DiBernardo showed an average skin surface area reduction of 22% and 17% at one- and three-month follow-up visits, respectively, and an average of 26% skin tightening at three months when utilizing LAL to address abdominal skin laxity<sup>20</sup>. In 2008, radiofrequency (RF) devices were introduced and have demonstrated efficacy in multiple body areas including the abdomen<sup>21,22</sup>, the arms<sup>23,24</sup>, and the face and neck<sup>25,26</sup>. The efficacy results in all of these publications are based on contraction measurements taken on the surface of the skin. Although skin surface contraction measurements are useful, they are limited for the following reasons:

- The mechanism of action (especially of Renuvion) is to treat and contract the fibro septal connective tissue. This contraction of the connective tissue draws the skin closer to the underlying muscle, and this, in turn, improves the appearance of the skin by reducing the laxity. When addressing skin laxity through the three-dimensional contraction of the connective tissue, the overall magnitude of improvement may not always be reflected in surface area changes on the skin surface. To date, no studies have measured the amount of contraction of the connective tissue itself.
- Using camera-based measurements of skin surface area changes do not allow for quantification of intraoperative (on the table) changes.
- Using camera-based measurements of skin surface area changes requires split-body treatments to differentiate between the results produced by liposuction and the energy device.

Due to these limitations, having another way to quantify and visualize contraction will be helpful. This study will use ultrasound images to visualize the contraction throughout the procedure and during follow-up. Utilizing those ultrasound images, this study will provide the ability to quantitatively measure the amount of soft tissue contraction produced by the delivery of Renuvion helium plasma energy to the subcutaneous connective tissue.

#### 2.1.1 Renuvion System Device and Indications for Use

The Renuvion APR system consists of a handpiece (Figure 1), an electrosurgical unit (ESU, Figure 2), and a supply of helium gas (Figure 2). RF energy is delivered to the handpiece by the ESU and used to energize an electrode. When helium gas is passed over the energized electrode, a helium plasma is generated which allows for conduction of the RF energy from the electrode to the subject in the form of a precise helium plasma beam.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol



FIGURE 1: RENUVION APR HANDPIECE



FIGURE 2: ELECTROSURGICAL UNIT AND HELIUM TANK

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

The Renuvion system has received FDA clearance under 510(k) numbers K223262 and K170188. The Renuvion® APR Handpiece is intended for the delivery of radiofrequency energy and/or helium plasma where coagulation/contraction of soft tissue is needed. Soft tissue includes subcutaneous tissue. The Renuvion® APR Handpiece is indicated for use in subcutaneous dermatological and aesthetic procedures to improve the appearance of lax (loose) skin in the neck and submental region. The Renuvion® APR Handpiece is intended to be used with compatible electrosurgical generators owned by Apyx Medical.

The Apyx One Console (K221830) is indicated for delivery of radiofrequency energy and/or helium plasma to cut, coagulate and ablate soft tissue during open and laparoscopic surgical procedures. The helium plasma portion of the generator can be used only with dedicated Renuvion/J-Plasma handpieces.

#### 2.1.1 ULTRASOUND SYSTEM AND INDICATIONS FOR USE

The GE Versana Active 1.5 (K200998) is a general-purpose diagnostic ultrasound system intended for use by qualified and trained healthcare professionals for ultrasound imaging, measurement, display and analysis of the human body and fluid. Versana Active clinical applications include: Fetal/Obstetrics, Abdominal, Gynecology, Urology, Pediatric, Small Organ (includes breast, testes, thyroid), Neonatal Cephalic, Adult Cephalic, Cardiac (includes Adult and Pediatric), Vascular/ Peripheral Vascular, Musculoskeletal Conventional, Musculoskeletal Superficial, Thoracic/ Pleural, Transcranial, Transrectal, Transvaginal, Interventional guidance (includes tissue biopsy, fluid drainage, vascular and non-vascular access). Modes of operation include: B, M, PW Doppler, CW Doppler, Color Doppler, Color M Doppler, Power Doppler, Harmonic Imaging, Coded Pulse, 3D, 4D and Combined modes: B/M, B/ Color M, B/PWD or CWD, B/Color/PWD or CWD, B/Power/PWD or CWD. The device is intended for use in an indoor hospital environment, in medical offices/clinics and other Healthcare facilities.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol



### 2.2 POTENTIAL RISKS AND BENEFITS

## 2.2.1 POTENTIAL RISKS

This treatment modality was designed to inherently minimize the risk to the subject. However, treatment with energy-based modalities (laser, radiofrequency, and plasma devices) produce subsequent heating of the soft tissue that could involve the following commonly Expected Treatment Effects (ETEs): discomfort/pain, edema, erythema, ecchymosis, hypoesthesia, temporary sensory nerve injury (touch sensitivity, itching, temporary numbness/tingling), transient migratory firmness, and temporary and/or transient crepitus.

In addition to commonly expected treatment effects, treatment with the Renuvion system could involve the following risks: helium embolism into the surgical site due to inadvertent introduction into the venous or arterial

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

blood supply system, unintended burns (deep or superficial), pneumothorax, temporary or permanent motor nerve injury, ischemia, fibrosis, infection, gas buildup, bleeding, hematoma, seroma, subcutaneous induration, pigmentation changes, increased healing time, unsatisfactory scarring, asymmetry and/or unacceptable cosmetic result.

Risks associated with tumescent anesthesia (lidocaine and epinephrine) include blurred vision, mental/mood changes, drowsiness, dizziness, unusually slow heartbeat, rash, itching, swelling, anxiety, apprehensiveness, restlessness, tremor, weakness, sweating, palpitations, pallor, nausea and vomiting, headache, and respiratory difficulties.

Subjects using drugs that reduce coagulation (aspirin or NSAIDs) may experience increased bruising or bleeding at the treatment site. Any other medication prescribed for the procedure or after-procedure by the investigator have their own risks; these risks should be discussed with the subject.

A grounding pad is used to ground/neutralize the electrical current. Subjects undergoing radiofrequency treatment will be kept away from contact with metal parts which are grounded, or which have appreciable capacitance to earth.

Any unexpected or unforeseen complications will be managed by the investigator throughout the conduct of the study. Unforeseen or unexpected side effects not listed above will be reported to the sponsor and regulatory representatives (IRB/EC) as they occur.

#### 2.2.1.1 MINIMIZATION OF POTENTIAL RISKS

These risks are mitigated by utilizing qualified clinical Investigators who have training and are experienced in procedures delivering radiofrequency energy and/or helium plasma where coagulation/contraction of soft tissue is needed and in the use of ultrasound systems. In addition, risks are mitigated by including only those subjects that meet the study eligibility criteria. This study also includes evaluation of study subject satisfaction with this procedure. Given the anticipated acceptable risk, the risk-benefit assessment of the use of the Renuvion APR device to deliver radiofrequency energy and/or helium plasma where coagulation/contraction of soft tissue is needed appears to offer a substantial clinical benefit at a reasonable risk.

#### 2.2.2 POTENTIAL BENEFITS

The benefit of this study is to add to the industry knowledge base a better understanding of the coagulation/contraction of soft tissue produced by the Renuvion APR system. Subjects enrolled in this study will receive the benefit of using the Renuvion APR device for the coagulation/contraction of soft tissue.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



## 3. STUDY PURPOSE

The purpose of this study is to quantitatively measure the amount of soft tissue contraction produced by the delivery of Renuvion helium plasma energy to the subcutaneous connective tissue.

## 4. STUDY DESIGN AND ENDPOINTS

## 4.1 DESCRIPTION OF THE STUDY DESIGN

This is a prospective, single-center, non-randomized study of up to 5 subjects who are receiving treatment with the Renuvion APR system following power-assisted liposuction in the abdomen per investigator standard of care. Subjects may also have other body areas treated at the same time. Demographic information, medical history, and procedure details will be documented. Pre- and post-procedure care are per investigator standard of care and documented. Video may be taken during the procedure.

Ultrasound images of soft tissue contraction will be taken on abdomen prior to and during the procedure. Measurements of contraction will be calculated from the ultrasound images by an ultrasonographer. At baseline, photographs will be taken of the treatment areas. Surface area measurements will be taken of each treatment area prior to study treatment.

Post-procedure care will be as per investigator standard of care and documented. All adverse events and expected treatment effects will be documented.

Follow-up photographs and ultrasound images will be captured at D30, D45, D60, D90, D180, D270, & D365.

An interim analysis of data will be completed following study treatments and following each follow-up visit (D30, D45, D60, D90, D180, D270); a final report will provide comprehensive study results through D365.

### 4.2 Duration of Study

Recruitment for this study may take approximately three (3) months. Following the treatment visit, subjects will be followed for a total duration of 365-days. Therefore, the anticipated total duration of the study is approximately sixteen (16) months.

#### 4.3 STUDY ENDPOINTS

#### 4.3.1 PRIMARY EFFECTIVENESS ENDPOINT

The primary effectiveness endpoint is an analysis of contraction measured by an ultrasonographer and then analyzed as follows:

- Quantify the amount of intra-operative contraction produced by liposuction.
- Quantify the amount of intra-operative contraction produced by each pass of Renuvion.
- Determine if amount of intra-operative contraction produced by Renuvion begins to level off (reach a point of diminishing return).
- Determine how the amount of intra-operative contraction varies based on the initial length at baseline.
- Correlate amount of intra-operative contraction to energy delivered.
- Determine how amount of contraction changes over time.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Correlate the amount of contraction to GAIS and PSQ.

- Correlate the amount of contraction or energy delivered to AEs.
- Correlate the amount of contraction to IPR review.

#### 4.3.2 SAFETY VARIABLES

The safety variables included in this study are as follows:

- Prior to treatment, the subject's medical history will be reviewed, a urine pregnancy test will be performed (if applicable), and a physical examination will be conducted.
- Following study treatment and at each subsequent visit, the subject will be queried about adverse events, expected treatment effects, and changes in concomitant medications, and the treatment area will be visually examined.
- Analysis of adverse events through the D365 post-treatment visit.

#### 4.3.3 Additional Outcome Measures

- 1. Improvement in appearance of skin laxity in the treatment area assessed by selection of the correct post-treatment image as determined by a masked, qualitative assessment of photographs by blinded independent reviewers at 90-days, 180-days, 270-days, and 365-days post-treatment compared to baseline.
- 2. The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a PGAIS assessing overall aesthetic improvement in the treatment area at day 60, 90, 180, 270, and 365 post-treatment.
- 3. The subject will complete a SGAIS assessing overall aesthetic improvement in the treatment area at day 60, 90, 180, 270, and 365 post-treatment.
- 4. The subject will complete a Patient Satisfaction Questionnaire (PSQ) at the 180-, 270- and 365-day follow-up visits.
- 5. Analysis of energy delivered per surface area and per volume of tissue.

#### 4.3.4 EVALUATION TOOLS

The following evaluation tools will be used in this study:

#### 4.3.4.1 Analysis of Contraction (Primary Outcome Measure)

Ultrasound images will be taken of the abdomen prior to and during the procedure, and at all follow-up visits. An experienced ultrasonographer will calculate the measurement of contraction. The measurements will be recorded on a study-specific Case Report Form (CRF). Measurements will be calculated as follows:

- Reproducible landmarks will be established on the ultrasound prior to beginning any treatment.
- The measurements will be taken from the underside of dermis to top of the muscle fascia.

Measurements will be calculated by the ultrasonographer at the following timepoints:

- At baseline (prior to any treatment before infiltration).
- Following liposuction.
- Following each Renuvion treatment pass.
- At all follow-up visits.

Utilizing the measurements calculated by the ultrasonographer, Apyx Medical or a contracted statistician will calculate the following contraction analyses:

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



- Quantification of the amount of intra-operative contraction produced by liposuction.
- Quantification of the amount of intra-operative contraction produced by each pass of Renuvion.
- Determine if amount of intra-operative contraction produced by Renuvion begins to level off (reach a point of diminishing return).
- Determine how the amount of intra-operative contraction varies based on the initial length at baseline.
- Correlate amount of intra-operative contraction to energy delivered.
- Determine how amount of contraction changes over time.
- Correlate the amount of contraction to GAIS and PSQ.
- Correlate the amount of contraction or energy delivered to AEs.
- Correlate the amount of contraction to IPR review.

#### 4.3.4.2 2-DIMENTIONAL PHOTOGRAPHY

Two-dimensional (2D) photographic images will be captured utilizing the study site's camera system. The same standardized views will be used throughout the study. Images will be taken at baseline, 30-day, 45-day, 60-day, 90-day, 180-day, 270-day, and 365-day visits.

#### 4.3.4.3 INDEPENDENT PHOTOGRAPHIC ASSESSMENTS

Three experienced, independent blinded photographic reviewers will perform a qualitative analysis/review of pretreatment and post-treatment sets of images for each subject. Images will be provided in a blinded and randomized order. Each blinded reviewer will choose which is the before image and which is the after. Success will be correct identification of before and after by at least 2 of the 3 reviewers.

#### 4.3.4.4 MODIFIED GLOBAL AESTHETIC IMPROVEMENT SCALE (GAIS)

The Modified Global Aesthetic Improvement Scale (GAIS) is a subjective rating of improvement in treatment results compared to pre-treatment. The Investigator will grade the overall improvement of abdominal treatment area as indicated in **Table 2** by comparing the subject's appearance at follow-up visits against a photograph taken prior to procedure. Likewise, the subject will also rate their improvement compared to pre-treatment as shown in **Table 3**.

The modified GAIS results will be collected at the 60-day, 90-day, 180-day, 270-day, and 365-day follow-up visits.

#### TABLE 3: MODIFIED GLOBAL AESTHETIC IMPROVEMENT SCALE EVALUATION - INVESTIGATOR

| Rating | Description |
|---|---|
| Very much improved | Optimal cosmetic result from this procedure in this subject |
| Much improved Marked improvement in appearance from the initial condition, but no completely optimal for this subject | |
| Improved | Obvious improvement in appearance from the initial condition |
| No change | ange The appearance is essentially the same as the original condition |
| Worse | rse The appearance is worse than the original condition |
| Much worse | uch worse The appearance is much worse than the original condition |
| Very much worse | ery much worse The appearance is very much worse than the original condition |

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 

| MEDICAL Apyx Medical Corporation | |
|---|---|
| Protocol Number: APX-23-02 | Effective Date: May 23, 2023 |
| Protocol Number: APX-23-02 | Revision No: 1.1 |
| Title: Measuring Renuyion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol | |

TABLE 4: MODIFIED GLOBAL AESTHETIC IMPROVEMENT SCALE EVALUATION - SUBJECT

| Rating |
|--------------------|
| Very much improved |
| Much improved |
| Improved |
| No change |
| Worse |
| Much worse |
| Very much worse |

Both scales should be completed in two steps:

- Based on a live assessment of the subject while referring to the subject's pre-treatment photographs (subjects should utilize a mirror for assessment); and
- Based on a comparison of the subject's pre-treatment photographs to the current post-treatment photographs.

#### 4.3.4.5 PATIENT SATISFACTION QUESTIONNAIRE (PSQ)

Patient Satisfaction Questionnaires (**Attachment B**) will be completed at the 180-day, 270-day, and 365-day follow-up visits. The subject should complete this assessment while referring to baseline photos, current photos, and a hand mirror.

#### 4.3.4.6 ADVERSE EVENT REPORTING

The definitions of Adverse Events (AEs) and the subtypes are provided in **Section 8** of the study protocol. Adverse events will be classified by the investigator as to:

- Serios vs not serious
- Expected Treatment Effect (ETE) vs Adverse Event (AE)
- Severity: mild, moderate, severe
- Device/procedure causality: not related, related, undetermined.

## 5. SUBJECT ENROLLMENT AND WITHDRAWAL

## 5.1 STUDY POPULATION

The study population will consist of males and females between 18 and 65 years of age who have chosen to participate in this clinical trial as evidenced by execution of the informed consent document and meet eligibility criteria defined in this protocol are eligible for participation in this clinical trial. Subjects will be considered enrolled into the study when they have signed an approved informed consent form. Subjects who are enrolled and do not meet eligibility criteria will be exited as a screen fail without study treatment. A study exit Case Report Form will be completed for all enrolled subjects.

#### 5.1.1 INFORMED CONSENT

Informed consent will be obtained from all subjects prior to study participation. Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. Extensive discussion of risks and possible benefits of participation will be provided to each participant.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

Investigators have ethical and legal responsibilities to ensure that the protocol is clearly explained to each subject considered for enrollment in the study. Compliance with this requirement should be documented on a written Informed Consent Form approved by the reviewing IRB. Each Informed Consent Form will include the elements required by FDA regulations in 21 CFR Part 50.

Consent forms will be IRB-approved, and the participant will be asked to read and review the document. The investigator, or investigator-delegated study personnel, will explain the research study to the participant and answer any questions that may arise. All participants will receive a verbal explanation in terms suited to their comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants will have the opportunity to carefully review the written consent form and ask questions prior to signing. The participants should have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The participant will sign the informed consent document prior to any procedures being done specifically for the study.

The IRB-approved Informed Consent Form will be signed by the study personnel obtaining consent. A copy of the informed consent document will be given to the participants for their records. The investigative site will keep the original on file. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

The participants may withdraw consent at any time throughout the course of the trial without any penalty or loss of benefits to which the subject is otherwise entitled. An Investigator may also discontinue a subject from the study without the subject's consent, if the Investigator feels it is in the best medical interest of the subject. The date and the reason for study withdrawal will be indicated on the Study Exit CRF.

#### 5.1.1.1 CONSENT/ASSENT AND OTHER INFORMATIONAL DOCUMENTS PROVIDED TO PARTICIPANTS

Consent forms describing in detail the study device, study procedures, and risks are given to the participant and written documentation of informed consent is required prior to starting intervention/administering study product.

#### 5.1.2 Pre-treatment Recruiting/Screening

Subjects will be recruited from the study site's patient database and social media and screened. Study site personnel will explain the design and purpose of the study to potential study subjects. Subjects interested in participating and who qualify will visit the study site where informed consent will be obtained. The site may utilize a pre-screening questionnaire that has been approved by the IRB.

### 5.1.2.1 SCREEN FAILURES

A screen failure subject is one from whom informed consent is obtained and is documented in writing (i.e., subject signs an Informed Consent Form), but who does not receive a study treatment because of failure to meet all of the eligibility criteria. Screen failure subjects will be included in the total number of subjects enrolled (i.e., all subjects consented), but not counted towards the total subjects treated.

#### 5.2 INCLUSION CRITERIA

Subjects must meet all of the following criteria for study enrollment:

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



- Patients who are scheduled for a procedure involving the use of Renuvion for the contraction of subcutaneous soft tissue. Patients undergoing procedures involving Renuvion following liposuction in the abdomen will be included.
- Patients who have acceptable cardiopulmonary health for outpatient surgery.
- Willing and able to comply with protocol requirements, including obtaining study-required images/photos and assessments, and returning for follow-up visits.
- Willing to release rights for the use of study photos, including in potential publication.
- Able to communicate with the site via video and/or photographs, in the event of a virtual follow-up visit.
- Able to read, understand, sign and date the informed consent document (English only).

#### 5.3 EXCLUSION CRITERIA

Subjects will be excluded if they meet any of the following criteria:

- BMI of greater than 35.
- Diabetes mellitus with A1C score >7.
- Active cigarette smokers or nicotine vape users.
- History of connective tissue disease (Ehlers Danlos, Cutis Laxa, Pseudoxanthoma Elasticum, Marfan's, etc.).
- Patients who, in the opinion of the investigator, are not an appropriate candidate for the study.
- Patients with a history of or requiring a concomitant procedure in the Renuvion treatment area that could impact the ultrasound measurements or the effectiveness results.

#### 5.4 STRATEGIES FOR RECRUITMENT AND RETENTION

Subjects will receive compensation for completion of the 30, 45, 90, 180, 270, and 365-day visits. This small stipend will be outlined in the site specific ICF and approved by the IRB prior to subject enrollment. The reason for the subject's withdrawal should be documented on the appropriate study specific CRF.

#### 5.5 Participant Withdrawal or Termination

#### 5.5.1 Reasons for Withdrawal or Termination

All subjects have the right to withdraw at any point during the study without prejudice. The investigator can discontinue any subject, at any time, if medically necessary. Subjects must be discontinued from the investigation by the investigator at any time for any of the following reasons:

- Withdrawal of informed consent.
- Pregnancy (no further study-related procedures will be performed).
- Any AEs for which treatment continuation would constitute an unacceptably high risk for the subject.

The reason for subject's withdrawal should be documented on the appropriate study specific CRF.

#### 5.5.2 HANDLING OF WITHDRAWALS OR TERMINATION

The subject must undergo the recommended follow-up assessments specified for the last study visit unless contraindicated due to a medical condition. Withdrawn subjects will not be replaced.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Effective Date: May 23, 2023

Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

Subjects who are discontinued from the study due to an AE(s) will be treated according to standard clinical practice and will be followed-up until the final study visit/safety visit. All pertinent information concerning the AE will be documented on the appropriate study specific CRF.

A subject may discontinue from the study at any time without any penalty or loss of benefits to which the subject is otherwise entitled. An Investigator may also discontinue a subject from the study without the subject's consent, if the Investigator feels it is in the best medical interest of the subject. The date and the reason for study withdrawal will be indicated on the Study Exit CRF.

#### 5.6 Premature Termination or Suspension of the Study or a Study Site

The study or a study site can be prematurely terminated or suspended by the sponsor. Reasons for termination of the study or a study site may include, but are not limited to, the following:

- Subject enrollment is unsatisfactory.
- The risks and benefits of continuing the study have been reassessed, and the risks outweigh any potential
- The incidence of AEs constitutes a potential health hazard to the subjects.
- New scientific data do not justify a continuation of the study.
- The investigator or study site exhibit serious and/or persistent non-adherence to the protocol, the Declaration of Helsinki, EN ISO 14155, and/or applicable regulatory requirements.
- The sponsor decides to terminate the study at any time for any other reason.

Furthermore, the study may be prematurely ended if the regulatory authority or the IRB has decided to terminate or suspend approval for the study, the study site, or the investigator.

If the study is prematurely terminated or suspended for any reason, the investigator must inform the subjects and assure appropriate follow-up treatment. Within the timeframes noted in applicable regulations, the sponsor will promptly inform the investigators, study sites, the IRB, and regulatory authorities of the termination or suspension of the study, as well as provide reasons for the action.

#### STUDY DEVICE 6.

Cleared Renuvion handpieces shipped for use in clinical investigations conform to the applicable general safety and performance requirements (GSPR) apart from the aspects covered by the clinical investigation and that, with regard to those aspects, every precaution is taken to protect the health and safety of the subjects. This includes, where appropriate, technical, and biological safety testing and pre-clinical evaluation as well as provisions in the field of occupational safety and accident prevention and taking into consideration the state of the art. Apyx Medical will provide Renuvion handpieces for use in this clinical investigation. The site will utilize their own Renuvion generator and ultrasound system.

#### 6.1 PACKAGING & STORAGE

The sponsor will provide appropriate packaging and storage instructions of the Renuvion handpieces to the study sites.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Effective Date: May 23, 2023

Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

#### 6.2 **ACCOUNTABILITY**

The investigator, or designee, must maintain an inventory record using the site-specific Device Disposition Form of study devices received, used for treatment, and returned to the Sponsor to ensure that the investigational device will not be dispensed to any person who is not a subject under the terms and conditions set forth in this protocol. There will be 100% accountability for all study devices. The clinical study site shall maintain all devices received for clinical trial use in a locked, limited access cabinet or room until the end of the study unless they are returned to Apyx while the study is being conducted, such as at the end of study treatments.

#### 6.3 Device Malfunction/Observation

All malfunctions of, or defects of the delivery system will be reported to the Sponsor by the study sites. This will include situations where the delivery system did not perform as intended; user errors; study device/component being physically defective, including out of the box failure.

#### 7. STUDY PROCEDURES AND SCHEDULE

#### 7.1 PRE-PROCEDURE

Study subjects will have verification of eligibility criteria, a brief general examination including medical history, and pre-procedure assessments as detailed below completed within 30 days prior to undergoing the study procedure. In response to the ongoing coronavirus disease (COVID-19) pandemic, preoperative testing can be completed at the Investigator's discretion. Pre-operative testing should be performed as close to the scheduled study procedure as feasible, but in time to get the results. Up to two urine pregnancy tests must be obtained prior to study procedure for females with child-bearing potential (one at pre-procedure screening and one on the day of the procedure prior to the procedure if pre-procedure screening and procedure are not performed on the same day).

The following pre-treatment assessments will be performed:

- 2D photographic images will be captured. The same standardized photography views will be used throughout the study.
- Urine pregnancy test (for females of childbearing potential).
- General physical exam including medical history, vital signs, collection of patient demographic information, and BMI.

Medications subject is taking upon entry into the study should also be documented in the Case Report Forms (CRF). All concomitant prescription medications taken during study participation will be recorded on the appropriate study specific CRF. For this protocol, a prescription medication is defined as a medication that can be prescribed only by a properly authorized/licensed clinician. Medications to be reported on the CRF and entered on the eCRF are concomitant prescription medications, over-the-counter medications, and non-prescription medications.

Medication used for analgesia and/or anesthesia should be recorded as concomitant medication as well. To ensure the capture of the foregoing information on pre-existing conditions, sites should also be attentive to the need to document without limitation and whenever discovered: (1) all chronic, episodic or 'as needed' medications used before study enrollment; (2) prior episodic or 'as needed' therapeutic interventions, procedures or hospitalizations; and, (3) recent or planned surgical procedures.

#### 7.2 STUDY PROCEDURE

On the day of the procedure and prior to the study procedure, female subjects with child-bearing potential must complete a urine pregnancy test (result must be obtained prior to the procedure), see Table 4.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

Medications at investigator discretion may be provided.

The abdominal procedure utilizing the Renuvion APR system will be performed per the investigator's standard clinical practice. Subjects may also have other body areas treated at the same time. Procedure data and adverse events will be captured.

Ultrasound Measurements of the abdomen will be collected intra-operatively (pre-treatment, post-liposuction, post each Renuvion pass). Video may be taken during the procedure.

#### 7.3 FOLLOW-UP PROCEDURES

#### 7.3.1 IMMEDIATELY POST-PROCEDURE

Following the procedure, the research staff and the subject will care for the treated areas using the Post-Procedure Care Instructions per the Investigator's standard clinical practice.

#### 7.3.2 FOLLOW-UP VISITS & SUBJECT CONTACT OUTSIDE OF FOLLOW-UP VISITS

The Investigator will follow-up with the study subjects per their Standard of Care (SOC), at the following time-points:

- 30 (±4) days
- 45 (±10) days
- 60 (±10) days
- 90 (±10) days
- 180 (±15) days
- 270 (±15) days
- 365 (±15) days

Post-procedure assessments, ultrasound imaging, and 2D photographic imaging will be performed during the follow-up visits, see **Table 4**. The same standardized photography views and ultrasound imaging will be used throughout the study as documented in the image capture document developed for the study.

Due to the challenges of COVID-19, if a subject is unable to return to the office for an in-person visit, follow-up visits will be conducted virtually. If a visit is completed virtually, missing assessments such as photographs will be documented as a protocol deviation specifically noting COVID-19. Outside of photographs, study investigators and study staff will ensure all other assessments related to each follow-up visit are completed virtually if the visit is done virtually. For virtual visits, the investigator and/or study staff completing the visit and assessments will be identified on the case report form; as well, the manner in which the visit was completed will also be recorded (i.e., video call, phone call, etc.). Virtual visits should be done via video call, if possible, to ensure subject identity. If a telephone call must be done, the investigator and/or study staff must positively identify the subject prior to conducting the virtual visit by requesting the subject to state their address and date of birth. Subjects will be strongly encouraged to come in (albeit safely) for their D365 visit; this visit is vitally important as this is the primary endpoint and photographic images are needed for many of the assessments. Only investigators and study staff who have been trained and delegated to conduct virtual visits as indicated on the delegation log may conduct virtual study visits.

Subjects may be seen for an unscheduled appointment at any time at investigator's discretion.

Study staff will contact (phone, text, email, video call at subject's preference) all subjects with ongoing Adverse Events at regular intervals. If the subject is unreachable by the preferred method of contact, another method of contact may be attempted.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

#### **TABLE 4: STUDY REQUIRED PROCEDURES**

| | Baseline/ Pre-<br>Procedure<br>Screening <sup>1</sup> | Procedure<br>(Day 0) | <b>30 Day</b><br>26-34<br>days | <b>45 Day</b><br>35-55<br>days | <b>60 Day</b><br>50-70<br>days | 90 Days<br>80-100<br>days | <b>180 Days</b><br>165-195<br>days | 270 Days<br>255-285<br>days | <b>365 Days</b><br>350-380<br>days |
|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | Х | | | | | | | | |
| Assess Inclusion/Exclusion Criteria | Х | | | | | | | | |
| Demographics | Х | | | | | | | | |
| Urine Pregnancy Test <sup>2</sup> | Х | Х | | | | | | | |
| Medical History | Х | | | | | | | | |
| General Physical Exam | Х | | | | | | | | |
| Review Medications | Х | х | Х | Х | Х | Х | Х | Х | Х |
| Photographic Imaging <sup>3</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Study Procedure | | Х | | | | | | | |
| Ultrasound<br>Imaging/Measurements <sup>4</sup> | | Х | Х | Х | Х | Х | Х | Х | x |
| Adverse Event Assessment | | Х | Х | Х | Х | Х | Х | Х | Х |
| Modified Global Aesthetic Improvement Scale (GAIS) <sup>5</sup> | | | | | Х | Х | Х | Х | х |
| Patient Satisfaction<br>Questionnaire <sup>6</sup> | | | | | | | Х | Х | х |

<sup>&</sup>lt;sup>1</sup> Pre-procedure Screening assessments to take place within 30 days prior to undergoing the procedure.

# 7.4 SUBJECT RANDOMIZATION AND TREATMENT GROUP ASSIGNMENT Subjects are not randomized in this study.

### 7.5 STUDY SCHEDULE

#### 7.5.1 Screening

- Obtain informed consent of potential participant verified by signature on study informed consent form.
- Verify all preliminary/screening inclusion/exclusion criteria are met.

## 7.5.2 BASELINE ASSESSMENT

- Document medical history.
- Obtain pregnancy screen (if applicable).
- Perform baseline photography.
- Document concurrent medications.
- Obtain height and weight.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 

<sup>&</sup>lt;sup>2</sup> Up to two urine pregnancy tests must be obtained prior to study procedure for females with child-bearing potential (one at pre-procedure screening and one on the day of the procedure prior to the procedure if screening and procedure are not performed on the same day).

<sup>&</sup>lt;sup>3</sup>Digital photographs will be taken and labeled according to Photography Instructions. Standard positioning and lighting will be used for all photographs.

<sup>&</sup>lt;sup>4</sup>To be taken intraoperatively (pre-treatment, post-liposuction, and post each Renuvion pass) and at each follow-up visit

<sup>&</sup>lt;sup>5</sup>To be completed by Investigator and study subject at day 60, day 90, day 180, day 270, and day 365 follow-up visits.

 $<sup>^6\</sup>mathrm{To}$  be completed by study subject at day 180, day 270, and day 365 follow-up visits.



Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

## 7.5.3 TREATMENT VISIT

- Greater than 30 days between baseline and treatment visits will require that the subject be re-screened to confirm enrollment eligibility.
- Obtain pregnancy screen (if applicable) prior to study treatment.
- Perform study treatment.
- Provide post-treatment instructions.

### 7.5.4 FOLLOW-UP

Subjects will be asked to return to the clinic for follow-up visits at 30-, 45-, 60-, 90-, 180-, 270-, and 365-days post-treatment. At all visits, subjects will be assessed for safety and efficacy, standardized images will be taken, ultrasound images will be taken for the independent ultrasonographer measurements, adverse events and protocol deviations will be assessed, and study outcome measures (GAIS, as applicable) will be completed. At the 180-day, 270-day, and 365-day follow-up appointment in addition to the above referenced assessments, the subject will complete a Patient Satisfaction Questionnaire.

#### 7.5.4.1 FOLLOW-UP ASSESSMENT AT 30+4 DAYS

- Obtain Images.
- Obtain ultrasound images for measurements.
- Assess/collect any adverse events.

#### 7.5.4.2 FOLLOW-UP ASSESSMENT AT 45+10 DAYS

- Obtain Images.
- Obtain ultrasound images for measurements.
- Assess/collect any adverse events

#### 7.5.4.3 FOLLOW-UP ASSESSMENT AT 60+10 DAYS

- Obtain Images.
- Obtain ultrasound images for measurements.
- Obtain aesthetic improvement scores.
- Assess/collect any adverse events

#### 7.5.4.3 FOLLOW-UP ASSESSMENT AT 90+10 DAYS

- Obtain Images.
- Obtain ultrasound images for measurements.
- Obtain aesthetic improvement scores.
- Assess/collect any adverse events.

#### 7.5.4.4 FOLLOW-UP ASSESSMENT AT 180+15 DAYS

- Obtain Images.
- Obtain ultrasound images for measurements.
- Obtain aesthetic improvement scores.
- Obtain patient satisfaction scores.
- Assess/collect any adverse events.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Effective Date: May 23, 2023

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

#### 7.5.4.5 FOLLOW-UP ASSESSMENT AT 270 +15 DAYS

- Obtain Images.
- Obtain ultrasound images for measurements.
- Obtain aesthetic improvement scores.
- Obtain patient satisfaction scores.
- Assess/collect any adverse events.

#### 7.5.4.6 FINAL VISIT AT 365 +15 DAYS

- Obtain Images.
- Obtain ultrasound measurements.
- Obtain aesthetic improvement scores.
- Obtain patient satisfaction scores.
- Assess/collect any adverse events.

#### 7.5.5 SAFETY ASSESSMENTS

Assess for adverse events immediately post-treatment and at all follow-up visits.

#### 7.5.6 Unscheduled Visit

Any unscheduled visit or examine should be documented in the subject's medical record and adverse event form (if applicable) stating the reason for the visit and any actions taken. The Sponsor should be notified of the unscheduled visit.

## 7.5.7 END OF STUDY (COMPLETION)

All subjects who have signed an Informed Consent Form will be considered enrolled in the study. Subjects who complete the study duration will be considered to have completed the study. The end of study will be defined as completion of all study visits by all enrolled subjects. If a device-related AE, SAE, or unanticipated serious devicerelated effect is ongoing at the final study visit, the subject will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or the subject is lost to follow-up.

A study closure visit may be conducted at the study site in order to review record retention requirements, device disposition requirements, etc., with site personnel. The Sponsor may choose to conduct the closure visit via telephone contact if appropriate.

#### ASSESSMENT OF SAFETY 8.

#### 8.1 Specifications of Safety Parameters

### DEFINITION OF AN EXPECTED TREATMENT EFFECT (ETE) AND AN ADVERSE EVENT (AE)

An expected treatment effect (ETE) is defined as any typical treatment side-effect of Renuvion APR of mild to moderate severity and lasting up to a typical maximum duration. An adverse event (AE) is defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject while enrolled in the study, whether or not it is considered device-related by the investigator.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Effective Date: May 23, 2023 Protocol Number: APX-23-02

Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

A preexisting condition (one that is present at the start of the study) will be recorded as an AE only if the frequency, intensity, or the character of the condition worsens during the study period. Neither the condition, hospitalization, prolonged hospitalization, nor surgery are reported as an AE in the following circumstances: hospitalization or prolonged hospitalization for diagnostic or elective surgical procedures for a preexisting condition. Surgery should not be reported as an outcome of an AE if the purpose of the surgery was elective or diagnostic and the outcome was uneventful.

All ETEs and AEs will be collected during the conduct of this trial.

### 8.1.2 Definition of Serious Adverse Event (SAE)

Each adverse event should be assessed for its seriousness. The definition below should be used for this assessment. Please note that the term serious adverse event is not synonymous with a "severe" adverse event, which may be used to describe the intensity of an event experienced by the subject.

An adverse event should be classified as serious if it meets any of the following criteria:

Death a.

Death was an outcome of the adverse event.

b. Life-threatening

The subject was at substantial risk of dying at the time of the adverse event or use or continued use of the device.

c. Hospitalization (initial or prolonged)

Admission to the hospital or prolongation of hospitalization was a result of the adverse event.

d. Disability or Permanent Damage

The adverse event resulted in a substantial disruption of a person's ability to conduct normal life functions, i.e., the adverse event resulted in a significant, persistent or permanent change, impairment, damage or disruption in the patient's body function/structure, physical activities and/or quality of life.

e. Congenital Anomaly/Birth Defect

Exposure to a medical product prior to conception or during pregnancy may have resulted in an adverse outcome in the child.

Required Intervention to Prevent Permanent Impairment or Damage (Devices)

Medical or surgical intervention was necessary to preclude permanent impairment of a body function, or prevent permanent damage to a body structure, either situation suspected to be due to the use of a medical product.

g. Other Serious (Important Medical Events)

The event does not fit the other outcomes, but the event may jeopardize the subject and may require medical or surgical intervention (treatment) to prevent one of the other outcomes.

Non-serious adverse events are all events that do not meet the criteria for a "serious" adverse event.

#### 8.1.3 Definition of Unanticipated Adverse Device Effects (Events)

An unanticipated adverse device effect is defined as "any serious adverse effect on health or safety, or any lifethreatening problem, or death caused by, or associated with, a device; if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, or application (including

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



supplementary application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects."

#### 8.2 Classification of an Event

#### 8.2.1 SEVERITY OF EVENT

Each adverse event should be assessed for its severity, or the intensity of an event experienced by the subject, using the following classifications:

- **Mild:** easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities. These events generally do not require treatment.
- **Moderate:** sufficiently discomforting to interfere with normal everyday activities. These events are usually relieved by simple therapeutic measures.
- **Severe:** prevents normal, everyday activities. These events may require systemic drug therapy or other medical treatment.

#### 8.2.2 Relationship to the Investigational Device

The **relationship to the study device and/or procedure** will be determined by the investigator utilizing the following categories:

- **Not Related:** An event for which an alternative explanation is conclusively identified e.g., concomitant drug(s), concomitant disease(s), and/or the relationship in time suggests that a causal relationship is highly unlikely.
- Related: The adverse event follows a reasonable temporal sequence related to treatment by the device and/or study procedure, follows a known or suspected response pattern and a plausible alternative etiology cannot be identified.
- **Undetermined:** The relation of the adverse event has some temporal relationship to the device and/or study procedure, is not clearly due to another condition and the involvement of the study device is unknown.

## 8.3 TIME PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP

The occurrence of an AE or SAE may come to the attention of study personnel during a study visit or upon review by a study monitor. All ETEs and AEs will be captured on the appropriate CRF. Information to be collected includes event description, date of onset, clinician's assessment of seriousness and severity, relationship to study device/treatment (assessed only by those with the training and authority to make a determination), actions taken, and date of event resolution. All AEs occurring while on study must be documented appropriately regardless of relationship. All device related ETEs/AEs assessed as "not yet resolved" must continue to be followed via telephone contact, email or clinic visit as per the physician's direction until event resolution or stabilization.

A pre-existing condition should not be reported as an adverse event unless there has been a substantial increase in severity or frequency of the problem that has not been attributed to natural history. Changes in the severity of an event will be documented to allow for a determination if the event should be re-categorized from an ETE to AE.

Safety evaluations for this study include an interview with the study subject at each follow-up visit by the Investigator or delegated study staff to elicit information about any medical occurrence that meets the definition of Adverse Event. This information will be documented in CRF without regard for cause or relation to device and/or procedure.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

Subjects may be asked by the study investigator to come into the site at any time to assess adverse events.

Study investigators are provided liberty to mitigate adverse events as deemed necessary per IHC GCP Guidelines E6(R2)4.3.2 which states "During and following a subject's participation in a trial, the investigator/institution should ensure that adequate medical care is provided to a subject for any adverse events related to the trial".

Adverse event resolution dates will be determined by investigator using either in-person or remote (phone, video call, text, email, etc.) examinations or communication with the subject. To ensure the most accurate reporting of adverse event durations, investigators are instructed not to wait until scheduled office follow-up visits to assess resolution.

It is the Investigator's responsibility to determine seriousness, severity, and relatedness of the Adverse Event to the device and procedure using the definitions in this protocol.

The PI will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of ETEs/AEs/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.

#### 8.4 REPORTING PROCEDURES

#### 8.4.1 Adverse Event Reporting

All Adverse Events (AEs) and Expected Treatment Effects (ETEs) observed by study subjects, investigators, or other study staff from first exposure to the study product through last study follow-up visit will be recorded. If a device-related AE, ETE, SAE, or unanticipated serious device related effect is ongoing at the final study visit, the subject will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or the subject is lost to follow-up. The investigator should make every effort to ensure that follow-up includes any supplemental investigations as may be indicated to elucidate, as completely as practical, the nature and/or causality of the AE or SAE. This may include unscheduled follow up visits for AE assessment.

Study subjects will be instructed in the ICF, post-treatment take home instructions, and verbally by study staff to report all AEs to the clinical study staff. AE information will be collected throughout the duration of the study and recorded on CRFs. Subjects experiencing ongoing adverse events will be contacted as per **Section 8.3**.

Any new medical problem, or an exacerbation of an existing condition, reported from the time the informed consent form is signed must be followed until the last study visit after the last study treatment or until event resolution.

AEs will not be followed up after the final study visit, which is scheduled <add time period in days, weeks or months> after the last study treatment.

#### 8.4.2 Serious Adverse Event Reporting

Serious adverse events must be reported to the Sponsor as soon as possible, preferably within 24 hours but in no event later than 72 hours. Any AE considered serious by the PI or Sub-investigator, or which meets the definition of an SAE included in **Definition of Serious Adverse Event** must be documented on an SAE CRF.

The Sponsor will conduct an investigation. If the Sponsor determines that the investigation presents an unreasonable risk to subjects, all investigations or parts of the investigation presenting that risk will be terminated as soon as possible. The investigator must report serious adverse events to the reviewing IRB/FDA according to the IRB/FDA regulations.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

#### 8.4.3 Unanticipated Adverse Device Effect Reporting

If an unanticipated adverse device effect occurs, the study investigator shall complete the appropriate study specific CRF and submit to the study sponsor and to the reviewing IRB as soon as possible, but in no event later than 10 working days after the investigator first learns of the effect. The study sponsor contact information is provided in **Apyx Medical Study Contact List**. The study sponsor is responsible for conducting an evaluation of an unanticipated adverse device effect and shall report the results of such evaluation to FDA and to all reviewing IRBs and participating investigators within 10 working days after the sponsor first receives notice of the effect. Thereafter the sponsor shall submit such additional reports concerning the effect as FDA requests.

#### 8.4.4 Reporting of Pregnancy

Each pregnancy that starts during the subject's study participation must be reported by the investigator to the Sponsor within 24 hours of learning of its occurrence. Pregnancies and pregnancy follow-up should be reported on an Adverse Event form. Pregnancy follow-up should describe the outcome of the pregnancy, including any voluntary or spontaneous discontinuation; details of the birth; the presence or absence of any congenital abnormalities, birth defects, maternal or newborn complications, and their relation to the device or treatment. Each pregnancy must be reported as a non-serious AE if the subject has received at least one study treatment. The following criteria should be followed:

- If a subject becomes pregnant after the Baseline visit and all study treatments have been completed, the subject should continue to be followed for the duration of the pregnancy.
- If a subject becomes pregnant after the Baseline visit but before any study treatments, the subject should be exited from the study.
- If a subject becomes pregnant after the Baseline visit but before all study treatments have been completed, additional study treatments should be discontinued, and the subject should continue to be followed for the duration of the pregnancy.

#### 8.4.5 Reporting of Deaths

The investigator must notify the Sponsor as soon as possible, preferably within 24 hours but in no event later than 48 hours, of learning of a subject's death, regardless of whether the death is related or unrelated to the investigational device. The investigator should attempt to determine, as conclusively as possible, whether the death is related to the device. The cause of death and the investigator's discussion regarding whether or not the death was device-related should be described in a written report. The investigator mush report death to the reviewing IRB according to the IRB regulations at the study site.

#### 8.5 STUDY HALTING RULES

This clinical trial will be halted if subjects' safety is questioned based on a reporting of severe, device-related AEs at an excessive frequency. The Sponsor and/or investigator may recommend termination or modification of the study if there is an occurrence of any device- or treatment-related Serious Adverse Event, using the clinical protocol definitions of Serious Adverse Event. In addition, termination or modification may be recommended for any other perceived safety concern based on clinical judgment, including but not limited to a severe burn (anticipated or unanticipated), a higher than anticipated rate for any component of the safety measures, device failures resulting in Adverse Events, or unexpected SAEs. The study sponsor will notify all investigators to immediately halt any continuing enrollment activities and not enroll any additional study participants. The study sponsor will inform the IRB/FDA of the temporary halt and the disposition of the study.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Effective Date: May 23, 2023

Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

The Sponsor and/or investigator may recommend termination or modification of the study if there is an occurrence of any device- or treatment-related Serious Adverse Event, using the clinical protocol definitions of Serious Adverse Event in Section 8.3 of this protocol. In addition, termination or modification may be recommended for any other perceived safety concern based on clinical judgment, including but not limited to a severe burn (anticipated or unanticipated), a higher than anticipated rate for any component of the safety measures, device failures resulting in Adverse Events, or unexpected SAEs. Enrollment and treatment would be suspended during root cause investigation to determine the cause of the respective AE.

#### **CLINICAL MONITORING** 9.

Clinical site monitoring is conducted to ensure that the rights and well-being of human subjects are protected, that the reported trial data are accurate, complete, and verifiable, and that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with applicable regulatory requirement(s). Details of clinical site monitoring are documented in the Study-specific Monitoring Plan (SMP), a separate document which documents in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level ofdetail monitoring will be performed, and the distribution of monitoring reports.

#### 10. STATISTICAL METHODOLOGY

#### 10.1 STATISTICAL AND ANALYTICAL PLANS

As this trial is exploratory in nature, not statistically powered, and has a very small sample size, only descriptive statistics will be used to summarize these data. Summarizes will include mean, standard deviation and median for continuous data and counts and frequencies for categorical data. 95% confidence intervals may be constructed, but it is recognized that they will be quite wide with such a small sample size.

#### 10.2 SAMPLE SIZE

The study will include up to 5 treated subjects from a single US site.

## SOURCE DOCUMENTS AND ACCESS TO SOURCE DATA/ 11. **DOCUMENTS**

Source documents are defined as the results of original observations and activities of a clinical investigation. Source documents will include, but are not limited to, study specific CRFs, progress notes, electronic data, computer printouts, screening logs, and recorded data from automated instruments. All source documents pertaining to this study will be maintained by the investigators and made available for inspection by authorized persons.

#### 12. QUALITY ASSURANCE AND QUALITY CONTROL

Quality Assurance and Quality Control procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution via data queries.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Effective Date: May 23, 2023

**Revision No: 1.1** 

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

Following written SOPs, the clinical study monitors will verify that the clinical trial is conducted, and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements.

The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

#### ETHICS/PROTECTION OF HUMAN SUBJECTS 13.

## 13.1 ETHICAL STANDARD

This clinical study will be conducted in accordance with the Protection of Human Subjects Regulations, including Subpart B Informed Consent of Human Subjects (21 CFR Part 50); the Institutional Review Board Regulations (21 CFR Part 56); the Financial Disclosure by Clinical Investigators Regulations (21 CFR Part 54); and the Investigational Device Exemptions Regulations (21 CRF Part 812), and the ICH E6 and in compliance with the Declaration of Helsinki, Council for International Organizations of Medical Science (CIOMS), International Ethical Guidelines for Biomedical Research Involving Human Subjects (2002), and EU MDR for protection of human subjects.

#### 13.2 Institutional Review Board

Prior to initiation of any study procedures, the protocol, informed consent, and recruitment materials, and all participant materials will be submitted to a duly constituted IRB for view and approval. In addition, any amendments to the protocol or Informed Consent Form will be reviewed and approved by the IRB. The Sponsor must receive a letter documenting IRB approval at the clinical site prior to the initiation of the study.

The investigator is responsible for providing the appropriate reports to its reviewing IRB during the course of the clinical study. These reports will include:

- Informing the IRB of the study progress periodically as required, but at least annually;
- Reporting any unanticipated adverse device effects within 10 working days of first learning of the event;
- Reporting any deviations from the clinical protocol to protect the life or well-being of a subject in the case of an emergency within five working days after the emergency occurred;
- Reporting the use of the device without obtaining informed consent from a subject within five working days of the event; and
- Providing any other reports requested by the IRB.

The IRB must be notified of study completion within 30 days of the final visit of the last subject and should be provided with a summary of the results of the study by the investigator.

#### PARTICIPANT AND DATA CONFIDENTIALITY

All information generated in this study must be considered highly confidential and must not be disclosed to any persons not directly concerned with the study without prior written permission from the Sponsor. Authorized regulatory officials and Sponsor personnel (or its representatives) will be allowed full access to inspect the records. Data disclosed outside the study team will be de-identified or will only include general group demographic

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

information. Protected Health Information and/or identifiable study data will not be shared with anyone outside the study team or Health System, with the exception of the study sponsor, and federal regulators/ institutional officials for the purposes of auditing.

All study devices and/or other materials collected will be used solely in accordance with this protocol, unless otherwise agreed to in writing by the Sponsor.

Subjects should be identified only by initials and unique subject numbers on study specific CRFs. If necessary, their full names may be made known to a regulatory agency or other authorized officials. Information to be stored on the computer will be identified by subject ID and will be password protected.

## DATA HANDLING AND RECORD KEEPING

#### 14.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site PI. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

During each subject's visit to the clinic, study data will be documented by study personnel on study-specific Case Report Forms (CRFs) prior to entry into an Electronic Data Capture (EDC) system. Subject demographic information, procedural data, adverse events, device observations, and study required assessments will be documented on the CRFs by delegated site personnel. Study subjects will complete Modified Global Aesthetic Improvement Scale (GAIS) Evaluations at protocol specified follow-up visits. Subjects will complete a Satisfaction Survey at the 60-day, 90-day, 180-day, 270-day, and 365-day follow-up visits. In addition, study personnel will record progress notes to document all significant observations, and any contact with a subject by telephone or other means that provides significant clinical information will also be documented in the progress notes as described above. In this clinical trial, study specific CRFs may serve as source documents.

For transmission to the Sponsor, information from the study progress notes and other source documents will be promptly transcribed to study specific CRF to the EDC with the CRF attached for remote monitoring of the data. Transcription of study data onto study specific CRFs and entry into the EDC should be completed within 3 days of the study visit.

Copies of the electronic CRF (eCRF) serving as source documents must be maintained for each participant enrolled in the study. Data reported in the eCRF derived from source documents should be consistent with the source documents or the discrepancies should be explained and captured in a progress note and maintained in the participant's official electronic study record.

Any changes to information in the study progress notes, other source documents, and CRFs will be initialed and dated in ink on the day the change is made by a site study staff member authorized to make the change. Changes will be made by striking a single line through erroneous data, and clearly entering the correct data. If the reason for the change is not apparent, a brief explanation for the change will be written in the source documentation by the investigator and/or delegated staff.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Photographic images will be captured utilizing the investigator's private practice camera system. Images will be uploaded to a secure site, Dropbox.com, for transfer to the study sponsor.

Data management and oversight is the responsibility of the Sponsor. A study specific Data Management Plan provides additional details.

Responsibilities may be delegated to applicable vendors.

#### 14.2 INVESTIGATOR RECORDS AND REPORTS

#### 14.2.1 INVESTIGATOR RECORDS

Prior to participation in the investigation, the investigator must provide the following documentation to the Sponsor:

- Investigator Agreement, signed by the investigator, which lists any physicians who will be involved in conducting the investigation under the direction of the primary investigator.
- A copy of the principal investigator's, sub-investigator's, other delegated study clinicians' curriculum vitae.
- A letter signed by the chairperson of the IRB overseeing the conduct of this study indicating that the IRB has reviewed and approved this investigational plan.
- A copy of the IRB-approved Informed Consent Form.

During the study, investigators are required to maintain on file the following accurate, complete, and current records relating to this study as described in 21 CFR §812.140. A summary of these records is listed below:

- Executed Clinical Trial Agreement.
- Signed Financial Disclosure.
- All correspondence and required reports, which pertain to the study, including IRB approvals and correspondence.
- Shipping documents and Device Disposition Log which records of receipt, use, or disposition of study devices, including the type and quantity of devices; the dates of receipt; the identifying product numbers; the names of all persons who received, used or disposed of each device; and why and how many units of the device have been returned to the Sponsor, repaired, or otherwise disposed.
- Records of each subject's case history and exposure to the device.
- Signed and dated consent forms.
- Relevant observations, including records concerning adverse events, condition of each subject upon entering and results of diagnostic tests.
- Study-specific CRFs and corrections to the forms.
- Protocol and amendments with signed Investigator Agreement/Statement of Compliance.
- IRB-approved subject recruiting materials.
- Investigator curriculum vitae and medical license.
- Monitoring reports and correspondence.
- Study logs including: Site Training Log, Site Visit Log, Site Delegation Log, and Subject Enrollment Log.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

#### 14.2.2 INVESTIGATOR REPORTS

Investigators are required to prepare and submit to the Sponsor the following complete, accurate, and timely reports on this investigation when are required. These reports, which are listed below, are required by 21 CFR §812.150; additional reports may be requested by the Sponsor:

- The investigator will notify the Sponsor of a subject death occurring during the investigation, as soon as possible, preferably within 24 hours of learning of the subject's death, but in no event later than 48 hours. The investigator will notify the reviewing IRB of a subject death as specified by the IRB.
- The investigator will notify the Sponsor of any unanticipated adverse device effects within 48 hours after learning of the effect. The investigator will notify its reviewing IRB of any unanticipated adverse device effects, as soon as possible, but no later than 10 working days after learning of the effect.
- The investigator will notify the Sponsor of the withdrawal of IRB approval, as soon as possible, but no later than five working days after learning of the withdrawal.
- The investigator will provide current progress reports to the Sponsor and reviewing IRB at regular intervals and at least on an annual basis.
- The investigator will notify the Sponsor and reviewing IRB of any deviation from the investigational plan to protect the life and physical well-being of a subject in an emergency, as soon as possible, but no later than five working days after the emergency occurred.
- The investigator will notify the Sponsor and reviewing IRB that an informed consent was not obtained from a subject, as soon as possible, but no later than five working days after such an occurrence.
- The investigator will provide a final summary report to the Sponsor and reviewing IRB within three months after termination or completion of the study.
- The investigator will provide any other information upon the request of an IRB, FDA, or the Sponsor.

## 14.3 STUDY RECORDS RETENTION

The investigator is responsible for retaining the necessary records, including a copy of the protocol, device labeling, study-specific CRFs, medical records, original reports of test results, all study-related correspondence, a record of written informed consent, and any other documents pertaining to the conduct of this study.

FDA regulations require all investigators participating in investigational device studies to maintain detailed clinical records during the investigation and for a period of at least two years after the latter of the following two dates:

- 1. The date on which the investigation is terminated or complete; or
- 2. The date the records are no longer required for purposes of supporting a premarket approval application.

The investigator must not dispose of any records relevant to this study without either:

- 1. Obtaining written permission from the Sponsor; or
- 2. Providing an opportunity for the Sponsor to collect such records.

The investigator shall take responsibility for maintaining adequate and accurate electronic or hard copy source documents of all observations and data generated during this study. Such documentation is subject to inspection by the Sponsor and the FDA.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

#### 14.4 PROTOCOL DEVIATIONS

A protocol deviation is an event in which the investigator or site personnel did not conduct the study in accordance with the protocol or the Clinical Trial Agreement. This study should be conducted as described in this protocol, except for an emergency situation in which the protection, safety, and well-being of a subject requires a protocol deviation, based on the judgment of the investigator (or a responsible, appropriately trained professional designated by the investigator). If the deviation from the protocol is necessary to protect the physical well-being of a subject in an emergency, such protocol deviations must be reported to the Sponsor and the reviewing IRB as soon as possible, but no later than five working days after the emergency occurred.

In the event of a significant deviation from the protocol due to an accident or mistake, the investigator or designee must contact the Sponsor at the earliest possible time to discuss the deviation and its impact on the study and subject continuation in the study. All protocol deviations and justification for the deviation will be documented on the applicable Case Report Form.

### 14.5 Publication and Data Sharing Policy

The data produced by this Apyx Medical-sponsored study is the sole property of Apyx Medical. Thereby, abstracts, publications and presentations of this data must be pre-approved by Apyx in writing (e-mail approval is acceptable). The Sponsor must also be provided with the opportunity to review all investigator-prepared abstracts, publications or presentations. A period of thirty (30) days for presentational materials and abstracts and forty-five (45) days for manuscripts will be required for review and comment by Sponsor's Clinical Affairs Department. These requirements acknowledge Sponsor's responsibility to evaluate such publications for their accuracy, to ascertain whether Confidential Information is being inappropriately released, to provide the Principal Investigator with information which may not yet have been available to him/her, and to provide input from co-authors regarding content and conclusions of the publication or presentation. If requested in writing by the Sponsor, the Institution will withhold publication to protect the potential patentability of any invention described therein and/or made available to fulfill regulatory requirements.

Notwithstanding the foregoing, Institution agrees that if the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results from the investigators at the other study centers as a multi-center publication.

The sponsor ensures that the study is registered, and study results are disclosed in at least one public clinical study registry, in accordance with national regulations and other requirements. Study registration may include a list of the study sites, as applicable.

## 15. STUDY ADMINISTRATION

## 15.1 STUDY INVESTIGATORS

Participating Investigators will be qualified based on professionals experienced in treatment delivering radiofrequency energy and/or helium plasma where coagulation/contraction of soft tissue is needed, such as plastic or cosmetic surgeons and the use of ultrasound systems. Investigators will be selected based on interest and availability for participation in the study; ability to provide qualified subjects; adequate support staff; experience conducting clinical research; and willingness to comply with the protocol, IRB requirements, regulatory requirements

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 



Effective Date: May 23, 2023 Protocol Number: APX-23-02

Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

(including the signed investigator agreement and statements disclosing any financial relationship investigators might have with Apyx Medical Corporation), and applicable regulations.

#### 15.2 **AMENDMENT POLICY**

The investigator will not make any changes to this protocol without prior written consent from the Sponsor and subsequent approval by the IRB, except if the deviation from the protocol is necessary to protect the life and physical well-being of a subject in an emergency. Such protocol deviations must be reported to the Sponsor and the reviewing IRB as soon as possible, but no later than five working days after the emergency occurred.

Any permanent change to the protocol, whether it is an overall change or a change for specific study center(s), must be handled as a protocol amendment. Any amendment to the protocol that appears indicated as the study progresses will be fully discussed by the investigator(s) and the Sponsor. If agreement is reached regarding the need for an amendment, the Sponsor will write it. The written amendment must be submitted to the chairman of the IRB identified with this responsibility. Except for "administrative amendments", investigators must await IRB approval of protocol amendments before implementing the change(s). Administrative amendments are defined to have no effect on the validity of the data or information resulting from the completion of the approved protocol, or the relationship of likely patient risk to benefit relied upon to approve the protocol; the scientific soundness of the investigational plan or protocol; and the right, safety or welfare of the human subjects involved in the investigation. When, in judgment of the chairman of the IRB, the investigators and/or the Sponsor, the amendment to the protocol substantially alters the study design and/or increases the potential risk to the subject, the currently approved written Informed Consent Form will require similar modification. In such cases, repeat informed consent will be obtained from subjects enrolled in the study before continued participation.

#### CONFLICT OF INTEREST POLICY 16.

The independence of this study from any actual or perceived influence is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the trial. The study leadership has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



Protocol Number: APX-23-02 Effective Date: May 23, 2023
Revision No: 1.1

Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol

## 17. LITERATURE REFERENCES

- 1. Feldman LS, Fuchshuber PR, Jones DB. The SAGES Manual on the Fundamental Use of Surgical Energy (FUSE). Springer Science+Business Media, LLC. 2012.
- 2. Goldberg SN, Gazelle GS, Halpern EF, Rittman WJ, Mueller PR, Rosenthal DI. Radiofrequency tissue ablation: importance of local temperature along the electrode tip exposure in determining lesion shape and size. Acad Radiol. 1996;3:212-8.
- 3. Thomsen S. Pathologic analysis of photothermal and photomechanical effects of laser-tissue interactions. Photochem Photobiol. 1991;53:825-35.
- 4. Ross EV, McKinlay JR, Anderson RR. Why does carbon dioxide resurfacing work? A review. Arch Dermatol 1999;135(4):444-454.
- 5. Gardner ES, Reinisch L, Stricklin GP, Ellis DL. In vitro changes in non-facial human skin following CO2 laser resurfacing: a comparison study. Lasers Surg Med 1996;19(4):379-387.
- 6. Doshi SN, Alster TS. Combination radiofrequency and diode laser for treatment of facial rhytides and skin laxity. Cosmet Laser Ther 2005;7:11-15.
- 7. Fatemi A, Weiss MA, Weiss RA. Short-term histologic effects of nonablative resurfacing: results with a dynamically cooled millisecond-domain 1320nm Nd:YAG laser. Dermatol Surg 2002;28(2):172-176.
- 8. Mayoral FA. Skin tightening with a combined unipolar and bipolar radiofrequency device. J Drugs Dermatol 2007;6(2):212-215.
- 9. Alster TS, Doshi SN, Hpping SB. Combination surgical lifting with ablative laser skin resurfacing of facial skin: a retrospective analysis. Dermatol Surg 2004;30(9):1191-1195.
- 10. Zelickson B, Kist D, Bernstein E, Brown DB, Ksenzenko S, Burns J, Kilmer S, Mehregan D, Pope K. Histological and ultrastructural evaluation of the effects of a radiofrequency-based nonablative dermal remodeling device: a pilot study. Arch Dermatol 2004;140:204-209.
- 11. Hsu T, Kaminer M. The use of nonablative radiofrequency technology to tighten the lower face and neck. Semin Cutan Med Surg 2003;22:115-123.
- 12. Paul M, Blugerman G, Kreindel M, Muholland RS. Three-dimensional radiofrequency tissue tightening: a proposed mechanism and applications for body contouring. Aesthetic Plast Surg. 2011;35(1):87-95.
- 13. Hurwitz D, Smith D. Treatment of overweight patients by radiofrequency-assisted liposuction (RFAL) for aesthetic reshaping and skin tightening. Aesthetic Plast Surg. 2012;36(1):62-71.
- 14. Duncan DI. Nonexcisional Tissue Tightening: Creating Skin Surface Area Reduction During Abdominal Liposuction by Adding Radiofrequency Heating. Aesthetic Surgery Journal. 2013;33(8):1154-1166.
- 15. Ulthera White Paper. Lower Face, Submentum, and Neck. Publicly available on <a href="www.ultherapy.com">www.ultherapy.com</a> by Ulthera Inc.
- 16. Boeni, R. Safety of Tumescent Liposuction under Local Anesthetsia in a Series of 4,380 Patients. Dermatology. 2011;222:278-281.
- 17. O'Brien Jr WD, O'Brien Jr WD. Assessing the risks for modern diagnostic ultrasound imaging. Japanese journal of applied physics. 1998 May 1;37(5S):2781.
- 18. Goldman A, Gotkin RH. (2009). Laser assisted lipolysis. Clin Plast Surg; 36(2):241-253.
- 19. Mordon S, Plot E. (2009). Laser lipolysis versus traditional liposuction for fat removal. *Expert Rev Med Devices*; 6(6):677-688.
- 20. DiBernardo BE, Reyes J. (2009). Evaluation of skin tightening after laser-assisted liposuction. *Aesthet Surg J;* 29(5):400–407. <a href="https://doi.org/10.1016/j.asj.2009.08.006">https://doi.org/10.1016/j.asj.2009.08.006</a>.
- 21. Duncan DI. (2013). Nonexcisional Tissue Tightening: Creating Skin Surface Area Reduction During Abdominal Liposuction by Adding Radiofrequency Heating. *Aesthet Surg J*; 33(8):1154-1166.
- 22. Paul M, Blugerman G, Kreindel M, Mulholland RS. (2011). Three-Dimensional Radiofrequency Tissue Tightening: A Proposed Mechanism and Applications for Body Contouring. *Aesth Plast Surg*; 35:87-95, doi:10.1007/s00266-010-9564-0

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



23. Duncan DI. (2012) Improving outcomes in upper arm liposuction: adding radiofrequency-assisted liposuction to induce skin contraction. *Aesthet Surg J*; 32(1):84-95, doi:10.1177/1090820X11429549. PMID: 22231416.

- 24. Chia CT, Theodorou SJ, Hoyos AE, Pitman GH. (2015). Radiofrequency-Assisted Liposuction Compared with Aggressive Superficial, Subdermal Liposuction of the Arms: A Bilateral Quantitative Comparison. *Plast Reconstr Surg Glob Open*; 3(7):e459. <a href="https://doi.org/10.1097/GOX.00000000000000429">doi:10.1097/GOX.0000000000000000429</a>. PMID: 26301148; PMCID: PMC4527633.
- 25. Key DJ. (2014). Integration of thermal imaging with subsurface radiofrequency thermistor heating for the purpose of skin tightening and contour improvement: a retrospective review of clinical efficacy. *J Drugs Dermatol*; 13(12):1485-9. PMID: 25607794.
- 26. Han X, Yang M, Yin B, Cai L, Jin S, Zhang X, Li F. (2021). The Efficacy and Safety of Subcutaneous Radiofrequency After Liposuction: A New Application for Face and Neck Skin Tightening. *Aesthet Surg J*; 41(3):NP94-NP100, doi:10.1093/asj/sjz364. PMID: 32004377.

Form-CLA-003-001 Title: Clinical Trial Protocol
Revision: 03 

| MEDICAL Apyx Medical Corporation | |
|---|---|
| Protocol Number: APX-23-02 | Effective Date: May 23, 2023 |
| Protocol Number: APX-23-02 | Revision No: 1.1 |
| Title: Measuring Renuvion Soft Tissue Contraction Using Ultrasound Clinical Trial Protocol | |

# ATTACHMENT A: PATIENT SATISFACTION QUESTIONNAIRE

Please have the subject complete this assessment while referring to their image in the mirror and current post-treatment photos compared to baseline photos. Provide the subject with a mirror.

Using a mirror and reviewing your post-treatment photos, compare how your treatment area currently looks compared to your pre-treatment photos.

| 1. | Do you notice ☐ YES → | ☐ Impro | ovement<br>sagging sk<br>other skin<br>e even ski | in wrinklo<br>kin<br>texture<br>n tone (co | es<br>olor) | domen lo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 2. | How would y Very Satis Satisfied Slightly S Slightly D Dissatisfie Very Diss | sfied<br>atisfied<br>satisfied o<br>vissatisfied<br>ed | r Dissatis | | action w | rith your p | rocedur | e? | | | |
| 3. | Would you re | ecommer | d this pro | | o your f | friends and | d family | member | s (check d | one)? | |
| 4. | On a scale fro | - | | | | - | - | erall sati | isfaction v | with the pro | ocedure and |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | Wors | t | | | | | | | | Best | |
| Thank y | ou for comple | eting this | question | naire. | | | | | | | |
| Subject | Initials: | | | Date | : | | | _ (DD/M | ON/YYYY | ") | |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 



# PROTOCOL REVISION LOG

**TABLE 5: PROTOCOL REVISION LOG** 

| VERSION | DATE | SIGNIFICANT REVISIONS |
|---------|-----------|------------------------------------|
| 1.0 | 4/21/23 | Initial Release |
| 1.2 | 5/23/2023 | Addition of Day 60 Follow-Up Visit |

Form-CLA-003-001 Title: Clinical Trial Protocol Revision: 03 